CLINICAL TRIAL: NCT05196789
Title: Diagnosis, Discovery and Novel Phenotype Characterisation Using Multimodal Genomics in Patients With Inherited Bone Marrow Failure and Related Disorders (IBMDx Study)
Brief Title: Diagnosis and Phenotype Characterisation Using Genomics in Patients With Inherited Bone Marrow Failure (IBMDx Study)
Acronym: IBMDx
Status: Recruiting | Type: Observational
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Other Study IDs: 77923
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Inherited BMF Syndrome; Inherited Platelet Disorder; Hematologic Diseases
Keywords: bone marrow failure syndrome; whole genome sequencing; hematological diseases; pancytopenia
MeSH Terms: conditions — Congenital Bone Marrow Failure Syndromes; Hematologic Diseases; Bone Marrow Failure Disorders; Pancytopenia | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, hair, skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: whole genome and transcriptome sequencing — To perform whole genome/transcriptome analysis of patients in a cohort of up to 350 Australian patients with IBMFS-RD

SUMMARY:
This project seeks to perform whole genome sequence (WGS) and whole transcriptome sequence (WTS) analysis on 350 patients with suspected inherited bone marrow failure syndromes and related disorder (IBMFS-RD) in order to increase the genomic diagnostic rate in IBMFS.

DETAILED DESCRIPTION:
IBMFS-RD are a heterogeneous group of rare diseases resulting in significant morbidity and early mortality. These syndromes are individually and collectively rare (affecting <1 per 10,000 people) and a significant proportion are unexplained by mutations in known genes. Whilst rare, these familial conditions are also likely underdiagnosed due to their relatively recent description and also due to lack of accessible genomic testing.

For patients with clinically suspected IBMFS-RD, receiving a genomic diagnosis is critical to:

* Establish a precise and reliable diagnosis (including distinguishing a monogenic aetiology from more common acquired or autoimmune causes of bone marrow failure which have dramatically different treatments (e.g. immunosuppression)
* Inform prognosis, clinical course, optimal treatment choice and screening for non-haematological organ dysfunction
* Optimise allogeneic haematopoietic stem cell transplant (HSCT) chemotherapy conditioning and minimise regimen-related toxicity
* Inform risk-benefit analysis of performing allogeneic HSCT to potentially prioritise other therapies (including novel gene therapy strategies)
* Avoiding the catastrophe of HSCT donation from occult genetically affected relatives
* Provide counselling (including stem cell donor counselling) and offer genetic testing for potentially affected family members
* Provide accurate reproductive counselling and reproductive options to affected individuals

This study aims to provide WGS and WTS to a national cohort of patients with IBMFS-RD to determine diagnostic rate, health economic impact, health implementation challenges and other exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 3 months
2. able to give informed consent (or parent/guardian able to give informed consent)
3. a clinicopathological diagnosis (or differential diagnosis) of inherited bone marrow failure syndrome or related disorder (IBMFS-RD) as per the study team

Exclusion Criteria:

1. A clinicopathological diagnosis of an acquired bone marrow failure syndrome (including acquired aplastic anaemia and hypoplastic myelodysplastic syndrome) as per the study team
2. Existing definitive genomic diagnosis for patient's haematological phenotype

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected IBMFS-RD
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Definitive IBMFS-RD diagnosis | 3-12 months post baseline
  IBMFS-RD diagnosis - An initial analysis of a panel of ~100 genes of established relevance to IBMFS-RD phenotype will be performed on all patients. If no molecular diagnosis is made from the panel of genes, further analysis on the genomic data will be performed using the best practice analytical tools and techniques.
  All results will be communicated to patients.

SECONDARY OUTCOMES:
Develop a whole transcriptome gene expression classifier | 4 years
  To develop a whole transcriptome gene expression classifier to aid diagnosis of IBMFS-RD.
Cost-effectiveness of genomic testing in patients with suspected IBMFS-RD | 4 years
  The cost-effectiveness of genomic testing is assessed by the differences in costs and quality of life associated with genomic testings compared with standard of care. Costs being considered include direct medical costs incurred within the health system arising from utilisation of hospital services and drug dispensing. Quality of life is assessed by EORTC-QLQ-C30 version 3 and CHU9D questionnaires for adult and paediatric patients respectively.
Budget-impact of genomic testing in patients with suspected IBMFS-RD | 4 years
  Evaluation of budget-impact of genomic testing includes examining the financial and operational sustainability as well as scalability of offering genomic testing beyond the trial period.
Health implementation analyses regarding the acceptability of genomic testing | 4 years
  The acceptability of comprehensive and centralised genomic testing in IBMFS-RD to patients is measured by a patient acceptability questionnaire which assesses patients' view and understanding of genomic testing.
Populate Registry | 4 years
  To populate the Aplastic Anaemia and Other Bone Marrow Failure Syndromes Registry (AAR, Monash University) with consenting patients with IBMFS-RD to facilitate long-term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Piers Blombery, MBBS(Hons), Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blombery P, Fox L, Ryland GL, Thompson ER, Lickiss J, McBean M, Yerneni S, Trainer A, Hughes D, Greenway A, Mechinaud F, Wood EM, Lieschke GJ, Szer J, Barbaro P, Roy J, Wight J, Lynch E, Martyn M, Gaff C, Ritchie D. Utility of clinical comprehensive genomic characterization for diagnostic categorization in patients presenting with hypocellular bone marrow failure syndromes. Haematologica. 2021 Jan 1;106(1):64-73. doi: 10.3324/haematol.2019.237693. PMID 32054657